CLINICAL TRIAL: NCT04539470
Title: A Phase Ib, Open-Label, Dose-Escalation Study to Evaluate the Safety and Pharmacokinetics of Efmarodocokin Alfa in Combination With Standard of Care in Patients Undergoing Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Study to Evaluate the Safety and Pharmacokinetics of Efmarodocokin Alfa in Combination With Standard of Care in Participants Undergoing Allogeneic Hematopoietic Stem Cell Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: GA41825
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Acute Graft-versus-host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A: Efmarodocokin Alfa Dosage Level 1 (Experimental): Participants undergoing allogeneic hematopoietic stem cell transplantation will receive Efmarodocokin Alfa dosage level 1 in combination with standard of care prophylaxis treatment for acute graft versus-host disease (aGVHD), consisting of tacrolimus plus methotrexate per institutional practices.
  Interventions: Drug: Efmarodocokin Alfa
- Cohort B: Efmarodocokin Alfa Dosage Level 2 (Experimental): Participants undergoing allogeneic hematopoietic stem cell transplantation will receive Efmarodocokin Alfa dosage level 2 in combination with standard of care prophylaxis treatment for acute graft versus-host disease (aGVHD), consisting of tacrolimus plus methotrexate per institutional practices.
  Interventions: Drug: Efmarodocokin Alfa
- Cohort C: Efmarodocokin Alfa Dosage Level 3 (Experimental): Participants undergoing allogeneic hematopoietic stem cell transplantation will receive Efmarodocokin Alfa dosage level 3 in combination with standard of care prophylaxis treatment for acute graft versus-host disease (aGVHD), consisting of tacrolimus plus methotrexate per institutional practices.
  Interventions: Drug: Efmarodocokin Alfa

INTERVENTIONS:
Drug: Efmarodocokin Alfa — Efmarodocokin Alfa will be administered intravenously (IV) per the dosage specified in each dose escalation cohort.
  Other Names: UTTR1147A; RG7880; RO7021610; IL-22Fc

SUMMARY:
This is a Phase Ib, open-label, multicenter, dose-escalation study to evaluate the safety, tolerability, and pharmacokinetics of Efmarodocokin Alfa and to make a preliminary assessment of activity of Efmarodocokin Alfa in combination with standard-of-care (SOC) in the prevention of acute graft-versus-host disease (aGVHD) in participants undergoing allogeneic hematopoietic stem cell transplantation (HSCT).

ELIGIBILITY:
Inclusion Criteria:

* Eligible for hematopoietic stem cell transplantation (HSCT)
* Donor meeting human leukocyte antigen (HLA) matching criteria of HLA-matched related or HLA-matched unrelated (HLA-A, HLA-B, HLA-C, and HLA-DRB1, eight out of eight) from either peripheral blood or bone marrow stem cells and meeting donor-eligibility criteria as outlined by the U.S. Food and Drug Administration (FDA) in 21 CFR 1271 (including screening for Zika and SARS-CoV-2 exposure or infection)
* Planned HLA (HLA-A, HLA-B, HLA-C, and HLA-DRB1)-matched (eight out of eight) related or planned HLA-matched (eight out of eight) unrelated HSCT, from either peripheral blood or bone marrow stem cells, for patients with acute myeloid leukemia (AML) or acute lymphocytic leukemia (ALL) in first complete remission (per institutional criteria) or patients with intermediate or high-risk myelodysplastic syndrome (MDS)
* Planned myeloablative conditioning regimen per institutional guidelines
* Planned aGvHD prophylaxis consisting of tacrolimus and methotrexate; in cases of tacrolimus intolerance, cyclosporine or sirolimus may be used as a substitute

Exclusion Criteria:

* Prior receipt of autologous or allogeneic HSCT
* Diagnosis of myelofibrosis or myelodysplastic/myeloproliferative overlap syndrome
* Treatment with investigational biologic or non-biologic therapy within 5 drug elimination half-lives (or within 90 days or 30 days, respectively, if half-life is unknown) prior to initiation of study drug
* Positive hepatitis B virus (HBV) or hepatitis C virus (HCV) serologies
* History of Grade >1 cervical intraepithelial neoplasia
* A marked baseline prolongation of QT/QTc interval
* Risk factors for torsades de pointes
* Pregnant or breastfeeding
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events by Severity, According to National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI-CTCAE v5.0) | From Baseline up to 365 days
Change from Baseline in Respiratory Rate Over Time | From Baseline up to 139 days
Change from Baseline in Oxygen Saturation Over Time | From Baseline up to 139 days
Change from Baseline in Pulse Rate Over Time | From Baseline up to 139 days
Change from Baseline in Systolic Blood Pressure Over Time | From Baseline up to 139 days
Change from Baseline in Diastolic Blood Pressure Over Time | From Baseline up to 139 days
Change from Baseline in Body Temperature Over Time | From Baseline up to 139 days
Number of Participants with Laboratory Abnormalities in Hematology Tests | From Baseline up to 139 days
Number of Participants with Laboratory Abnormalities in Blood Chemistry Tests | From Baseline up to 139 days

SECONDARY OUTCOMES:
Serum Concentration of Efmarodocokin Alfa at Specified Timepoints | At predefined timepoints from Baseline until Day 139
Number of Participants with Anti-Drug Antibodies (ADAs) at Baseline and During the Study | At predefined timepoints from Baseline until Day 139

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (8):
- United States (8):
  - City of Hope, Duarte, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - University of Miami Miller School of Medicine; Clinical Reseach Building, Miami, Florida
  - University of Chicago, Chicago, Illinois
  - University of Kansas Med Ctr; Int med/Allgy/Immun/Rheum, Kansas City, Kansas
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to individual patient level data through the request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/).
  For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).